CLINICAL TRIAL: NCT00003053
Title: Adjuvant Treatment of Non Small Cell Lung Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Stage I, II, or IIIA Non-small Cell Lung Cancer That Has Been Surgically Removed
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Institute of Oncology (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065700; CNR-NICO-01; EU-97010
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2008-01

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Etoposide; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: cisplatin
Drug: etoposide
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare cisplatin and etoposide with no chemotherapy in treating patients who have stage I, stage II, or stage IIIA non-small cell lung cancer that has been surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the efficacy of the combination of cisplatin and etoposide after radical surgery in prolonging the relapse free and overall survival for stages I, II, and IIIA non-small cell lung cancer.

OUTLINE: This a randomized study (treatment vs no treatment). Patients are stratified according to sex and to stage of disease (I vs II vs IIIA).

Patient receives cisplatin and etoposide on days 1-3, every 28 days, for 3 cycles. Patient may receive radiation therapy after surgery at the discretion of the physician.

PROJECTED ACCRUAL: Approximately 750 patients will be accrued over 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage I, II, or IIIA non-small cell lung cancer after radical surgery
* No evidence of lymphonodal enlargement during postsurgical chest CT scan

PATIENT CHARACTERISTICS:

Age:

* 70 and under

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Not specified

Renal:

* Creatinine no greater than 1.5 times the upper limit of normal

Pulmonary:

* FEV1 at least 1 liter

Other:

* Less than 10% weight loss in the past 3 months
* No prior malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Radical surgery required

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 1994-01

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Nicolucci, MD, Study Chair — Consorzio Mario Negri Sud
Locations (86):
- George Papanicolaou General Hospital, Thessaloniki, Greece
- Italy (84):
  - Ospedale Bassini, Balsamo Cinisello
  - Universita Degli Studi di Bari Policlinico, Bari
  - Spedali Civili, Brescia
  - Ospedale Oncologico A. Businco, Cagliari
  - Cattedra di Oncologia Medica - Universita degli Studi di Cagliari, Cagliari
  - Ospedale San Michele, Cagliari
  - Ospedale Sant Anna, Como
  - Ospedale Valduce, Como
  - Ospedale Di Conselice, Conselice
  - Ospedale Civile Cosenza, Cosenza
  - Ospedale Maggiore Crema, Crema
  - Ospedale Santa Croce, Cuneo
  - Ospedale Civile Feltre, Feltre
  - Universita di Ferrara, Ferrara
  - Universita Degli Studi di Firenze - Policlin. di Careggi, Firenze (Florence)
  - Policlinico di Careggi, Firenze (Florence)
  - U.S.L. 10 Villa Ognissanti, Florence
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa (Genova)
  - Ospedale San Martino/Cliniche Universitarie Convenzionate, Genoa (Genova)
  - Ospedale Galliera Oncologia, Genova (Genoa)
  - Ospedale Di Gorgonzola, Gorgonzola
  - Ospedale Alessandro Manzoni, Lecco
  - Ospedale Legnago USSL 21, Legnago
  - Ospedale Maggiore Lodi, Lodi
  - Ospedale Umberto I, Lugo DI Romagna
  - U.S.S.L. 72 Magenta, Magenta
  - Carlo Poma Hospital, Mantova
  - Ospedale Di Predabissi Melegnano, Melegnano
  - Azienda USSL NO 8, Merate
  - Instituto Di Oncologia, Messina
  - Ospedale Civile Umberto I, Mestre
  - Ospedale San Giuseppe, Milan
  - Consorzio Provinciale Antitubercolare, Milan
  - Istituto Scientifico H.San Raffaele, Milan
  - Istituto Di Science Biomediche San Paolo, Milan
  - Casa Di Cura San Ambrogio, Milan
  - Ospedale San Carlo Borromeo, Milano (Milan)
  - Ospedale Luigi Sacco, Milano (Milan)
  - Ospedale Maggiore Ca'Granda, Milano (Milan)
  - Ospedale Santa Croce, Moncalieri
  - Nuovo Ospedale San Gerardo, Monza
  - Ospedale Civile Asilo Vittoria, Mortara
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples
  - Federico II University Medical School, Naples (Napoli)
  - Istituto Tumori/Fondazione Pascale, Naples (Napoli)
  - Ospedale Vincenzo Monaldi, Napoli
  - Ospedale C. Ascalesi, Napoli
  - Ospedale Civile Negrar, Negrar
  - Azienda Ospedaliera di Padova, Padova (Padua)
  - University of Padua, Padua
  - Ospedale Civico E Benefratelli, Palermo
  - Ospedale Maggiore Parma, Parma
  - Ospedale Torrette University Ancona, Parma
  - Ospedale Silvestrini, Perugia
  - Ospedale Agnelli, Pinerolo
  - Ospedale Sta. Maria Delle Croci, Ravenna
  - Azienda Ospedaliera, Reggio Emilia
  - Ospedale Civile Rho, Rho
  - Istituti Fisioterapici Ospitalieri - Roma, Rome
  - Ospedale San Filippo Neri, Rome
  - Ospedale Carlo Forlanini, Rome
  - Ospedale S. Camillo-Forlanini, Rome
  - Azienda Policlinico Umberto Primo, Rome
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
  - Policlinico Militare Celio, Rome
  - ASL NO. 1 Imperiese, Sanremo
  - Consorzio Mario Negri Sud, Santa Maria Imbaro
  - Azienda USSL No 4, Saronno
  - Istituto Clinica Medica, Sassari
  - Ospedale Sesto San Giovanni, Sesto San Giovanni
  - Azienda Ospedaliera S. Maria, Terni
  - Ospedale Generale Prov. Boldrini, Thiene
  - Dispensario Igiene Sociale, Toino
  - Clinica Universita, Torino
  - Universita di Torino, Torino
  - Ospedale S. Chiara, Trento
  - Ospedale San Isidoro, Trescore Balneario
  - Ospedale General Regional Ca Foncello, Treviso
  - Ospedale Maggiore dell' Universita, Trieste
  - Ospedale Cattinara, Trieste
  - Cattedra di Immunologia Clinica, Turin (TO)
  - Universita Degli Studi di Udine, Udine
  - Casa di Cura S. Maria, Varese
  - Ospedale San Bortolo, Vicenza
- Inha University Hospital, Incheon, South Korea